CLINICAL TRIAL: NCT07121998
Title: Longitudinal Biomarker Study in Endocrine Neoplasms to Study Acquired Resistance to Alkylator Chemotherapy
Brief Title: Study of Acquired Resistance to Alkylator Chemotherapy in Endocrine Neoplasms
Acronym: PROGRESS-TMZ
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Joakim Crona, Associate professor, Clinical oncologist, Uppsala University Hospital
Other Study IDs: V1.1
Record Dates: First submitted 2025-06-17; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Neuroendocrine (NE) Tumors; Endocrine Cancer
Keywords: Alkylating chemotherapy; Treatment resistance
MeSH Terms: conditions — Neoplasms; Endocrine Gland Neoplasms | interventions — Biopsy, Large-Core Needle; Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with endocrine neoplasms who have or will receive treatment with alkylating chemotherapy.: Group A (about to start alkylating chemotherapy) Group B (at progression, previous alkylating chemotherapy)
  Interventions: Procedure: Core needle biopsy; Procedure: Phlebotomy

INTERVENTIONS:
Procedure: Core needle biopsy — Core needle biopsy of metastatic lesions
Procedure: Phlebotomy — Phlebotomy of peripheral vein

SUMMARY:
It has been showed that alkylating chemotherapy, particularly the widely used agent temozolomide, may cause high tumor mutational burden (TMB) in certain tumors by causing inactivating mutations in the DNA mismatch repair (MMR) system. This can cause therapy resistance and tumor progression but may also predict response for immunotherapy. Hypermutation is very uncommon in neuroendocrine tumors. However, small studies indicate that around 30% of pancreatic tumors develop high TMB after alkylating chemotherapy. The aim of this study is therefore to study the occurrence and frequency of DNA hypermutation after alkylating chemotherapy in endocrine neoplasms and to investigate non-invasive methods that may capture the development of hypermutation (imaging, ctDNA etc.).

This is a prospective multicenter study. 94 patients from Swedish endocrine cancer centers in Uppsala, Stockholm, Göteborg and Lund will be included and divided into two groups. Group A will include patients that are about to start treatment with alkylating chemotherapy. Blood samples for liquid biopsy will be collected at baseline and at follow-up and if the tumor progresses, tissue biopsy will be obtained from two different lesions and analyzed with GMS560. Group B will include patients experiencing tumor progression after having received alkylating chemotherapy at any point in their disease course before. At inclusion, both liquid and tissue biopsy will be obtained and analyzed as described above.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age ≥18 years
* Histopathology confirmed endocrine neoplasm
* Treatment with alkylating chemotherapy: Arm A; about to start alkylating chemotherapy, or Arm B; at disease progression or recurrence with previous alkylating chemotherapy treatment.

Exclusion Criteria:

* If planned tissue biopsy: risk factors for biopsy-related complications accordingly to local investigator, including coagulation disorder
* Long term treatment with anticoagulant that cannot be temporarily paused without unacceptable risk
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with endocrine neoplasms who have or will receive treatment with alkylating chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of pancreatic neuroendocrine tumor patients with hypermutation and/or mismatch repair deficiency after treatment with alkylating chemotherapy | Through study completion, an average of 2 years.
  Proportion of pancreatic neuroendocrine tumor patients with hypermutation (tumour mutation burden >30) and/or mismatch repair deficiency (by DNA sequencing or immunohistochemistry) in tissue or liquid biopsy at any timepoint after treatment with alkylating chemotherapy.

OTHER OUTCOMES:
Proportion of non-pancreatic endocrine neoplasms that develop hypermutation and/or mismatch repair deficiency after treatment with alkylating chemotherapy | Through study completion, an average of 2 years.
  Do non-pancreatic endocrine neoplasms (adrenocortical carcinoma, pheochromocytoma and paraganglioma, lung carcinoids and intestinal neuroendocrine tumors) develop hypermutation (tumor mutation burden >30) and/or mismatch repair deficiency (by DNA sequencing or immunohistochemistry) in tissue or liquid biopsy at any timepoint after treatment with alkylating chemotherapy?

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Crona, MD PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Akademiska Sjukhuset, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No